CLINICAL TRIAL: NCT07159386
Title: Metabolic Dysfunction-associated Steatotic Liver Disease (MASLD) in Primary Care
Brief Title: Advanced Fibrosis Detection for MASLD in Primary Care
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Andrew Schreiner, Associate Professor-Faculty, Medical University of South Carolina
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: Pro00145783
Record Dates: First submitted 2025-08-05; First posted 2025-09-08 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Metabolic Dysfunction-associated Steatotic Liver Disease
Keywords: Diabetes; Liver; Obesity
MeSH Terms: conditions — Diabetes Mellitus; Obesity

STUDY DESIGN:
Intervention Model Description: Study design: A stepped-wedge, cluster randomized clinical trial with an open cohort design using convergent, parallel mixed-methods to study: (i) the detection of advanced fibrosis in patients with known MASLD; and (ii) the implementation of a non-interruptive EHR alert for MASLD fibrosis risk assessment in primary care. All outcomes will be compared between unexposed (control) and exposed (intervention) periods.
  Randomization and Blinding: All clinics will begin the study in the control phase. The intervention will be introduced in 5 steps with 5-6 clinics per step at intervals of 6 months. The transition phase from the control period to the intervention period will last 1 month and provide time for rolling out educational content and access to the EHR alert. A computer-generated randomization program will assign clinics to one of the 5 pre-defined transition steps (months 6, 12, 18, 24, and 30).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Month 6 (Experimental): All clinics will begin the study in the control phase. The intervention will be introduced in 5 steps with 5-6 clinics per step at intervals of 6 months. The transition phase from the control period to the intervention period will last 1 month and provide time for rolling out educational content and access to the MASLD fibrosis risk assessment EHR alert. A computer-generated randomization program will assign clinics to one of the 5 pre-defined transition steps (months 6, 12, 18, 24, and 30).
  Interventions: Other: EHR alert
- Month 12 (Experimental): All clinics will begin the study in the control phase. The intervention will be introduced in 5 steps with 5-6 clinics per step at intervals of 6 months. The transition phase from the control period to the intervention period will last 1 month and provide time for rolling out educational content and access to the MASLD fibrosis risk assessment EHR alert. A computer-generated randomization program will assign clinics to one of the 5 pre-defined transition steps (months 6, 12, 18, 24, and 30).
  Interventions: Other: EHR alert
- Month 18 (Experimental): All clinics will begin the study in the control phase. The intervention will be introduced in 5 steps with 5-6 clinics per step at intervals of 6 months. The transition phase from the control period to the intervention period will last 1 month and provide time for rolling out educational content and access to the MASLD fibrosis risk assessment EHR alert. A computer-generated randomization program will assign clinics to one of the 5 pre-defined transition steps (months 6, 12, 18, 24, and 30).
  Interventions: Other: EHR alert
- Month 24 (Experimental): All clinics will begin the study in the control phase. The intervention will be introduced in 5 steps with 5-6 clinics per step at intervals of 6 months. The transition phase from the control period to the intervention period will last 1 month and provide time for rolling out educational content and access to the MASLD fibrosis risk assessment EHR alert. A computer-generated randomization program will assign clinics to one of the 5 pre-defined transition steps (months 6, 12, 18, 24, and 30).
  Interventions: Other: EHR alert
- Month 30 (Experimental): All clinics will begin the study in the control phase. The intervention will be introduced in 5 steps with 5-6 clinics per step at intervals of 6 months. The transition phase from the control period to the intervention period will last 1 month and provide time for rolling out educational content and access to the MASLD fibrosis risk assessment EHR alert. A computer-generated randomization program will assign clinics to one of the 5 pre-defined transition steps (months 6, 12, 18, 24, and 30).
  Interventions: Other: EHR alert

INTERVENTIONS:
Other: EHR alert — Diagnoses of MASLD (based on ICD 9/10 code) in a patient's EHR history, visit, or problem list, will cue a non-interruptive alert to appear and prompt clinicians to use the integrated EPIC© FIB-4 calculation SmartPhrase. The tool displays the FIB-4 risk score, the advanced fibrosis risk, and the clinical guidance. LSM by ultrasound with elastography will be recommended for patients with FIB-4 >1.3 (FIB-4 >2.0 if age >65) and the decision support will urge clinicians to order US with elastography through the SmartSet. LSM results will be documented in the EHR and categorized as low-risk MASLD (LSM <8 kPa) or advanced fibrosis (LSM >8 kPa). Results will be disseminated to the ordering PCPs and the patients. PCPs will receive information on patient counseling for MASLD, and the expanding roles of weight loss, reduced alcohol use, and exercise on disease management. PCPs will be encouraged to refer patients with advanced fibrosis to a hepatology specialist, in accordance with guidelines.

SUMMARY:
This proposal evaluates the implementation of a novel, non-interruptive, electronic health record alert for metabolic dysfunction-associated steatotic liver disease (MASLD) fibrosis risk assessment in primary care patients with MASLD using a stepped wedge, cluster randomized design. This work will generate generalizable data to dramatically enhance MASLD management in primary care.

DETAILED DESCRIPTION:
Metabolic dysfunction-associated steatotic liver disease (MASLD, formerly nonalcoholic fatty liver disease [NAFLD]) affects an estimated 1in 3 persons in the U.S., a prevalence expected to increase over the next decade. MASLD's rising prevalence and its association with diabetes and obesity make it a chronic disease well-suited for initial management by primary care providers (PCPs). PCPs can impact MASLD care by first detecting advanced fibrosis, which is the best predictor of cirrhosis, hepatocellular carcinoma, and liver-related mortality in affected patients. Recently issued guidelines from the American Association for the Study of Liver Diseases recommend the sequential use of non-invasive liver tests, the Fibrosis-4 Index (FIB-4) followed by confirmatory liver stiffness measurement (LSM) with vibration-controlled elastography (VCTE), to detect advanced fibrosis in patients with MASLD. FIB-4 is attractive in primary care due to the low-cost and broad availability of its inputs, but PCPs have little experience with FIB-4 calculation, limited comfort with its interpretation, and infrequent access to confirmatory liver stiffness testing. The guidelines provide a clinical threshold for hepatology engagement, recommending referral for patients with advanced fibrosis, while those with low-risk MASLD remain in primary care. Incorporating advanced fibrosis detection into the already overwhelming workload of PCPs requires thoughtful application of electronic health record (EHR)technologies to avoid contributing to PCP alert fatigue and burnout. In this work, investigators aim to evaluate the adoption, penetration, fidelity, sustainability, and performance of a novel, non-interruptive EHR alert for MASLD fibrosis risk assessment in a primary care network by performing a stepped wedge, cluster randomized trial in patients with known or suspected MASLD (Aim 1). This proposal aligns with NIDDK's scientific goal to disseminate, implement, and evaluate evidence-based care strategies in community care settings where the burden of MASLD hides in plain sight.

ELIGIBILITY:
Patients

Inclusion Criteria:

* Patients with a diagnosis code for MASLD
* Type 2 diabetes mellitus will

Exclusion Criteria:

* All patients with cirrhosis, complications of cirrhosis (e.g. portal hypertension, hepatic encephalopathy), hepatocellular carcinoma, or previous liver transplant will be excluded.
* pregnant women.

Clinicians Clinicians will also be study participants, as we will be surveying them for feedback on the MASLD fibrosis risk assessment intervention. The MUSC primary care network at last count employed 122 clinicians across the 27 primary care practices.

Inclusion criteria:

1. All physicians, physician assistants, and nurse practitioners delivering primary care during the intervention phase of the study.

Exclusion criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2030-09 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Detection of advanced fibrosis | Up to five years after implementation of the intervention.
  The primary clinical outcome of interest is the detection of advanced fibrosis. This outcome will be determined by reviewing US with elastography results from the medical record. Advanced fibrosis will be categorized by LSM >8 kPa (no advanced fibrosis is LSM <8 kPa)

SECONDARY OUTCOMES:
Implementation Adoption: Percentage of eligible MASLD patients who receive an order for liver stiffness testing. | Up to five years after implementation of the intervention.
  For the implementation outcomes, we will measure the adoption of the MASLD care intervention. We will quantify this outcomes using Proctor's implementation outcomes framework.
Implementation Penetration: Percentage of PCPs who order liver stiffness testing for eligible MASLD patients. | Up to five years after implementation of the intervention.
  We will measure the penetration of the MASLD care intervention. We will quantify this outcomes using Proctor's implementation outcomes framework.
Implementation Fidelity: Percentage of eligible MASLD patients who complete liver stiffness testing after receiving an order. | Up to five years after implementation of the intervention.
  We will measure the fidelity, and sustainability of the MASLD care intervention. We will quantify this outcomes using Proctor's implementation outcomes framework.
Implementation Sustainability: Percentage of clinics maintaining use of the MASLD fibrosis risk assessment alert over time. | Up to five years after implementation of the intervention.
  We will measure the sustainability of the MASLD care intervention. We will quantify this outcomes using Proctor's implementation outcomes framework.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Schreiner, MD, MSCR, Principal Investigator — Medical University of South Carolina

IPD SHARING:
Plan to Share IPD: No
Data will be used internally for implementation evaluation and quality improvement.